CLINICAL TRIAL: NCT06941116
Title: Steroids-Based Screening for Primary Aldosteronism
Acronym: SAFE
Status: Recruiting | Type: Observational
Sponsor: Qifu Li (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Chief Physician, Department of Endocrinology, The First Affiliated Hospital of Chongqing Medical University., Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: SAFE Study
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: Steroid-Based Screening; Aldosterone-to-Renin Ratio (ARR); Machine Learning; Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples will be retained. Plasma samples collected at multiple time points will be stored at -80°C for subsequent steroid hormone and biochemical analyses. Urine samples collected randomly during the standardized screening visit will also be stored at -80°C for further biochemical assessment. No samples will be used for DNA extraction or genetic analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PA Group: Participants with confirmed primary aldosteronism (PA)
  Interventions: Diagnostic Test: Steroid-Based Screening (LC-MS/MS)
- EH Group: Participants with essential hypertension (EH)
  Interventions: Diagnostic Test: Steroid-Based Screening (LC-MS/MS)

INTERVENTIONS:
Diagnostic Test: Steroid-Based Screening (LC-MS/MS) — This diagnostic intervention is a liquid chromatography-tandem mass spectrometry (LC-MS/MS)-based steroid profiling assay. It measures a panel of 18 adrenal steroid hormones (e.g., aldosterone, 18-hydroxycortisol, 18-oxocortisol, corticosterone) from plasma samples. In this study, it is used to screen for Primary Aldosteronism (PA) while patients remain on their usual antihypertensive medications. By comparing these steroid profiles against standard aldosterone-renin measurements, the method aims to reduce the need for medication washout and improve diagnostic accuracy for PA.

SUMMARY:
This prospective, single-center observational study aims to evaluate whether a steroid-based screening method can more accurately identify Primary Aldosteronism (PA) in hypertensive patients who remain on their usual antihypertensive medications, compared with the conventional aldosterone-to-renin ratio (ARR). PA is a common, potentially curable subtype of secondary hypertension that carries increased cardiovascular risk when undiagnosed or untreated. However, current screening protocols recommend "medication washout" or switching to minimally interfering drugs, which may pose safety concerns and add complexity.

In this study, approximately 406 participants (ages 18-75) with diagnosed hypertension and on at least one interfering antihypertensive drug (such as ACE inhibitors, ARBs, beta-blockers, diuretics, or calcium channel blockers) will be enrolled at the Department of Endocrinology, The First Affiliated Hospital of Chongqing Medical University. Each participant will undergo two rounds of blood sampling-first while continuing their usual antihypertensive regimen (the "on-medication" state) and second following a standardized washout/switch period (the "standard state"), if medically feasible. At both stages, levels of plasma aldosterone, renin, and a broad panel of adrenal steroid hormones will be measured by liquid chromatography-tandem mass spectrometry.

By comparing diagnostic performance (e.g., sensitivity, specificity, and area under the receiver operating characteristic curve) of the steroid-based screening versus the ARR, the study seeks to determine whether steroid profiling improves accuracy under real-world treatment conditions. Findings may help refine PA screening strategies, reduce the need for extensive medication adjustments, and contribute to better clinical management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, with no sex restriction.
2. Diagnosed with hypertension, defined as a systolic blood pressure ≥140 mmHg and/or a diastolic blood pressure ≥90 mmHg measured on at least two different days.
3. Currently receiving at least one antihypertensive medication that interferes with aldosterone or renin (ACEI/ARB, β-blockers, dihydropyridine CCBs, or diuretics including MRA) for ≥4 consecutive weeks.
4. Fully informed about the study procedures and risks, and willing to participate by signing a written informed consent form.

Exclusion Criteria:

1. Confirmed secondary hypertension of other etiologies (e.g., renovascular hypertension, renal artery stenosis, reninoma, pheochromocytoma, Cushing's syndrome, Liddle syndrome), excluding obstructive sleep apnea.
2. Severe cardiac, hepatic, or renal impairment or serious infections, including but not limited to New York Heart Association (NYHA) Class III-IV heart failure, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels exceeding 2.5 times the upper limit of normal, estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m², or severe infections (e.g., diabetic foot, sepsis, pneumonia, refractory infections).
3. History of major cardiovascular or cerebrovascular events within the past 3 months.
4. Pregnant or breastfeeding women.
5. Currently using medications (other than the listed antihypertensives) that may affect aldosterone or renin secretion, including but not limited to sex hormones (e.g., oral contraceptives, estrogen replacement therapy), glucocorticoids (e.g., prednisone, dexamethasone), nonsteroidal anti-inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen), or antipsychotics (e.g., chlorpromazine, olanzapine).
6. Individuals lacking or having restricted capacity for independent decision-making or action.
7. History of psychiatric disorders.
8. Poor compliance likely to compromise study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients diagnosed with hypertension (aged 18-75) who are receiving at least one antihypertensive medication that interferes with aldosterone or renin. Participants are recruited from the Endocrinology Outpatient Clinic at The First Affiliated Hospital of Chongqing Medical University between April 2025 and December 2026. All candidates must meet the predefined inclusion criteria (e.g., on interfering antihypertensive drugs for ≥4 weeks) and provide written informed consent. Patients with other confirmed forms of secondary hypertension or severe comorbidities are excluded. The anticipated sample size is approximately 406 participants.
Sampling Method: Non-Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Steroid-Based Screening vs. ARR for Primary Aldosteronism in Patients on Antihypertensive Medications | From baseline screening while on medication to completion of confirmatory testing, approximately 4-8 weeks.
  The primary outcome is to compare the diagnostic accuracy (e.g., sensitivity, specificity, area under the ROC curve [AUC]) of a steroid-based screening approach with the conventional aldosterone-to-renin ratio (ARR) for identifying primary aldosteronism (PA) in participants who remain on interfering antihypertensive medications (ACE inhibitors, ARBs, beta-blockers, diuretics, or calcium channel blockers). Confirmatory tests (e.g., captopril challenge, saline infusion) in a standard (washed-out) state will be used as the reference standard. A higher AUC or better sensitivity/specificity indicates superior performance.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, MD, PhD, Chief Physician, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We do not intend to share individual participant data from this study due to concerns regarding participant privacy, regulatory constraints, and the limited scope of the current study. Aggregated or summary results will be made publicly available through publication or the results section on ClinicalTrials.gov.

REFERENCES:
- [Background] Constantinescu G, Gruber S, Fuld S, Peitzsch M, Schulze M, Remde H, Kurzinger L, Yang J, Yen T, Williams TA, Muller L, Reincke M, Lenders JWM, Beuschlein F, Pamporaki C, Eisenhofer GF. Steroidomics-Based Screening for Primary Aldosteronism: Impact of antihypertensive Drugs. Hypertension. 2024 Oct;81(10):2060-2071. doi: 10.1161/HYPERTENSIONAHA.124.23029. Epub 2024 Jul 31. PMID 39082132
- [Background] Eisenhofer G, Duran C, Cannistraci CV, Peitzsch M, Williams TA, Riester A, Burrello J, Buffolo F, Prejbisz A, Beuschlein F, Januszewicz A, Mulatero P, Lenders JWM, Reincke M. Use of Steroid Profiling Combined With Machine Learning for Identification and Subtype Classification in Primary Aldosteronism. JAMA Netw Open. 2020 Sep 1;3(9):e2016209. doi: 10.1001/jamanetworkopen.2020.16209. PMID 32990741
- [Background] Li X, Liang J, Hu J, Ma L, Yang J, Zhang A, Jing Y, Song Y, Yang Y, Feng Z, Du Z, Wang Y, Luo T, He W, Shu X, Yang S, Li Q; Chongqing Primary Aldosteronism Study (CONPASS) Group. Screening for primary aldosteronism on and off interfering medications. Endocrine. 2024 Jan;83(1):178-187. doi: 10.1007/s12020-023-03520-6. Epub 2023 Oct 5. PMID 37796417
- [Background] Liu X, Hao S, Bian J, Lou Y, Zhang H, Wu H, Cai J, Ma W. Performance of Aldosterone-to-renin Ratio Before Washout of Antihypertensive Drugs in Screening of Primary Aldosteronism. J Clin Endocrinol Metab. 2024 Nov 18;109(12):e2302-e2308. doi: 10.1210/clinem/dgae094. PMID 38381080
- [Background] Fischer E, Beuschlein F, Bidlingmaier M, Reincke M. Commentary on the Endocrine Society Practice Guidelines: Consequences of adjustment of antihypertensive medication in screening of primary aldosteronism. Rev Endocr Metab Disord. 2011 Mar;12(1):43-8. doi: 10.1007/s11154-011-9163-7. PMID 21331645
- [Background] Mulatero P, Monticone S, Deinum J, Amar L, Prejbisz A, Zennaro MC, Beuschlein F, Rossi GP, Nishikawa T, Morganti A, Seccia TM, Lin YH, Fallo F, Widimsky J. Genetics, prevalence, screening and confirmation of primary aldosteronism: a position statement and consensus of the Working Group on Endocrine Hypertension of The European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1919-1928. doi: 10.1097/HJH.0000000000002510. PMID 32890264
- [Background] Griffin TP, Browne GA, Wall D, Dennedy MC, O'Shea PM. A cross-sectional study of the effects of beta-blocker therapy on the interpretation of the aldosterone/renin ratio: can dosing regimen predict effect? J Hypertens. 2016 Feb;34(2):307-15. doi: 10.1097/HJH.0000000000000775. PMID 26867057
- [Background] Browne GA, Griffin TP, O'Shea PM, Dennedy MC. beta-Blocker withdrawal is preferable for accurate interpretation of the aldosterone-renin ratio in chronically treated hypertension. Clin Endocrinol (Oxf). 2016 Mar;84(3):325-31. doi: 10.1111/cen.12882. Epub 2015 Sep 22. PMID 26300226
- [Background] Mulatero P, Rabbia F, Milan A, Paglieri C, Morello F, Chiandussi L, Veglio F. Drug effects on aldosterone/plasma renin activity ratio in primary aldosteronism. Hypertension. 2002 Dec;40(6):897-902. doi: 10.1161/01.hyp.0000038478.59760.41. PMID 12468576
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Background] Calhoun DA, Nishizaka MK, Zaman MA, Thakkar RB, Weissmann P. Hyperaldosteronism among black and white subjects with resistant hypertension. Hypertension. 2002 Dec;40(6):892-6. doi: 10.1161/01.hyp.0000040261.30455.b6. PMID 12468575
- [Background] Brown JM, Siddiqui M, Calhoun DA, Carey RM, Hopkins PN, Williams GH, Vaidya A. The Unrecognized Prevalence of Primary Aldosteronism: A Cross-sectional Study. Ann Intern Med. 2020 Jul 7;173(1):10-20. doi: 10.7326/M20-0065. Epub 2020 May 26. PMID 32449886
- [Background] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Background] Choy KW, Fuller PJ, Russell G, Li Q, Leenaerts M, Yang J. Primary aldosteronism. BMJ. 2022 Apr 20;377:e065250. doi: 10.1136/bmj-2021-065250. No abstract available. PMID 35443988